CLINICAL TRIAL: NCT04100356
Title: The Effect of Exercise and/or Diet Body Composition, Cardiorespiratory Fitness and Blood Parameters Related to Improved Health in Overweight Females.
Brief Title: The Effect of Exercise and/or Diet on Health Related Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantis Medical University College (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: AMUC-NIH-LCHF-P3-2014
Record Dates: First submitted 2019-09-13; First posted 2019-09-24 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Overweight and Obesity
Keywords: Low-carbohydrate-high-fat diet (LCHF); Low-density-lipoprotein (LDL); High-density-lipoprotein (HDL); Triglycerides (TG); Lipids; Glucose tolerance (GT); Insulin resistance (IR); Body composition; Weight
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Body Weight | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Diet and exercise, or diet only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal diet (Experimental): The group ingests normal diet, recommended by the health authorities
  Interventions: Other: Normal Diet
- LCHF diet (Experimental): The group ingests LCHF diet, a modified Atkins diet with 70 energy percentage fat
  Interventions: Other: LCHF Diet
- Normal diet + exercise (Experimental): The group ingests normal diet, recommended by the health authorities in addition to exercise program 3x week.
  Interventions: Other: Exercise; Other: Normal Diet
- LCHF diet + exercise (Experimental): The group ingests LCHF diet, a modified Atkins diet with 70 energy percentage fat, in addition to exercise program 3x week.
  Interventions: Other: Exercise; Other: LCHF Diet

INTERVENTIONS:
Other: Exercise — Exercise program - indoor bicycle interval exercise, duration 60 min 3x week
  Arms: LCHF diet + exercise; Normal diet + exercise
Other: Normal Diet — Normal diet recommended by the health authorities
  Arms: Normal diet; Normal diet + exercise
Other: LCHF Diet — LCHF Diet, a modified Atkins diet with high percentage of fat and very low percentage of karbohydrates
  Arms: LCHF diet; LCHF diet + exercise

SUMMARY:
The study evaluates the effect of exercise and/or diet during on body weight, body composition and health related blood parameters. Participants are overweight sedentary females, allocated to four different groups: Normal diet, Low-carb-high-fat diet, Normal diet + exercise, Low-carb-high-fat diet + exercise.

DETAILED DESCRIPTION:
Diet and exercise can both be efficient tools to reduce bodyweight, get healthier body composition and improve many different health related blood parameters such as cholesterol and glucose tolerance.

Exercise has superior effect on skeletal muscle in the context of glucose tolerance, but adherence to exercise program can be a huge challenge for overweight individuals. While exercise has profound effect on metabolic health, diet has been superior when it comes to weight reduction. Previous studies have shown that 5-7% weight loss can improve glucose tolerance, measured as reduced fasting glucose and reduced 2-hour post prandial glucose.

We wish to see if the combination exercise and diet is superior to diet only when it comes to over all health.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Sedentary
* Premenopausal
* Caucasian
* BMI 26.9 - 36.1
* Age 33-4
* Living close to, or in Oslo.

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Smoking or tobacco use
* Previous medical history of cardio-vascular disease (CVD)
* Previous medical history of diabetes
* Previous medical history of endocrine disorder
* Previous medical history of kidney disease
* Use of lipid lowering medication
* Use of diabetes medication

Ages: 33 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Premenopausal
Enrollment: 57 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2014-04-04 (Actual); Study Completion 2014-04-23 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) glucose | Change from baseline AUC glucose at 10 weeks
  AUC glucose measured during an OGTT

SECONDARY OUTCOMES:
Lipid profile | Change from Baseline lipids at 10 weeks
  Measurements of total cholesterol, LDL, HDL, TG
Body composition | Change from baseline values at 10 weeks
  Measurement of lean body mass, fat free mass, fat mass, visceral fat, bone mass
Cardiorespiratory fitness | Change from baseline values at 10 weeks
  Measurement of peak oxygen uptake

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Jensen, Professor, Principal Investigator — Norwegian School of Sport Sciences, Section of Physical Performance
Locations (1):
- Norwegian School of Sports Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valsdottir TD, Ovrebo B, Kornfeldt TM, Litleskare S, Johansen EI, Henriksen C, Jensen J. Effect of aerobic exercise and low-carbohydrate high-fat diet on glucose tolerance and android/gynoid fat in overweight/obese women: A randomized controlled trial. Front Physiol. 2023 Jan 24;14:1056296. doi: 10.3389/fphys.2023.1056296. eCollection 2023. PMID 36760521